CLINICAL TRIAL: NCT02855060
Title: Pre-hospital Advanced Therapies for Control of Hemorrhage (PATCH) - Pelvis
Brief Title: Pre-hospital Advanced Therapies for Control of Hemorrhage - Pelvis
Acronym: PATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-15-08B
Record Dates: First submitted 2016-07-27; First posted 2016-08-04 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-07

CONDITIONS: Hemorrhage; Pelvic Fracture
MeSH Terms: conditions — Hemorrhage; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelvic Binder (Experimental): Commercially available device used to stabilize the pelvis
  Interventions: Device: Pelvic Binder
- No Binder (No Intervention): Standard of care

INTERVENTIONS:
Device: Pelvic Binder
  Arms: Pelvic Binder

SUMMARY:
The purpose of this study is to determine whether the use of pelvic binders in the ambulance setting improves outcomes including mortality in patients with pelvic fractures.

DETAILED DESCRIPTION:
The goal of this prospective, randomized clinical trial is to determine whether prehospital use of a commercial pelvic binder will improve morbidity and mortality in patients with pelvic fractures. We hypothesize that prehospital placement of pelvic binders will reduce hemorrhage and need for resuscitation and will improve overall mortality in patients with pelvic fractures. In addition, we hypothesize that pelvic splinting via external compression will improve patients' pain regardless of whether they have a pelvic, acetabular, or proximal femur fracture.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic injury other than ground-level fall, and
* Complaint of pelvic groin or hip pain, or
* Pelvic or hip deformity, ecchymosis, or crepitus in an obtunded patient, or
* Hemodynamic instability

Exclusion Criteria:

* Ground level fall
* Penetrating pelvis injury without frank evidence of fracture
* Obviously pregnant patients
* Patients who are too small or too big for the binder
* Priority 2 or 3 Trauma

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pelvic Binder: Commercially available device used to stabilize the pelvis
  Pelvic Binder
Period: Overall Study
Arm/Group | Pelvic Binder | No Binder
Started | 22 | 28
Completed | 20 | 23
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pelvic Binder | No Binder | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.5 [27.0 to 45.0] | 36.0 [24.0 to 49.0] | 36.0 [26.0 to 47.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rate
Description: Percentage of patients that experience mortality within 30 days of presentation will be compared between the two study arms
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Binder | No Binder
Number analyzed (Participants) | 20 | 23
Participants | 0 | 1

2. Secondary Outcome: Pain Scores - Visual Analog Scale
Description: Pain scores at presentation to hospital will be compared between the two study arms. Range 0-10. Higher scores indicate a worse outcome.
Time Frame: At time of arrival to Emergency Department
Population: Pain scores were not documented in the Emergency Department for all patients. Only patients with scores documented were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pelvic Binder | No Binder
Number analyzed (Participants) | 12 | 15
score on a scale | 8.5 [7.5 to 10] | 10.0 [7.0 to 10.0]

3. Secondary Outcome: Number of Participants With Skin Complications After Pelvic Binder Application
Description: The rate of occurrence of skin complications after binder application will be documented.
Time Frame: From date of randomization to date of discharge or date of death from any cause, whichever came first, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Binder
Number analyzed (Participants) | 20
Participants | 0

4. Secondary Outcome: Length of Stay in Hospital
Description: The total number of days the patient spent in the hospital
Time Frame: From date of admission to date of discharge or date of death from any cause, whichever came first, assessed up to 1 year
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pelvic Binder | No Binder
Number analyzed (Participants) | 20 | 23
days | 3.0 [0 to 10] | 7.5 [2.5 to 16.5]

5. Secondary Outcome: Number of Patients With Blood Transfusions
Description: Number of Blood Transfusions within the first 48 hours after hospital admission
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Binder | No Binder
Number analyzed (Participants) | 20 | 23
Participants | 1 | 5

ADVERSE EVENTS:
Time Frame: 30 day
Description: Medical record was reviewed for all patients after 30 days
Arm/Group | Pelvic Binder | No Binder
All-Cause Mortality (participants affected / at risk) | 0/22 | 2/28
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/28
Other Adverse Events (participants affected / at risk) | 0/22 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02855060/Prot_SAP_000.pdf